CLINICAL TRIAL: NCT06153901
Title: Metal Clip and Endoloop Mediated Endoscopic Cardioplication (ECLC) for the Treatment of Gastroesophageal Reflux Disease (GERD):a Prospective Cohort Study
Brief Title: Endoloop Mediated Cardioplication to Treat Gastroesophageal Reflux Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Shandong University (Other)
Responsible Party: Principal Investigator, Lu Jiaoyang, professor, Qilu Hospital of Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-QILU-LU 02
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Gastroesophageal Reflux Disease; Endoscopy Upper GI Tract; anti-reflux; Endoscopic therapy
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- endoloop mediated cardioplication (ECLC) (Experimental): The ECLC surgery first incises the mucosa and submucosa on the small curvature side and posterior side (approximately 3/4 of the total circumference) of the diaphragm level cardia until smooth muscle fibers are exposed; Fix the metal clip covered with nylon rope on the exposed smooth muscle layer, and finally tighten the nylon rope to achieve full folding of the cardia. After the surgery, the patient fasted overnight and received intravenous PPI treatment. On the second day after surgery, a fluid diet was restored and discharge was possible. ECLC is simple, easy to operate, relatively inexpensive, and minimally invasive, and is expected to become a new method for treating severe gastroesophageal reflux disease.
  Interventions: Procedure: endoloop mediated cardioplication (ECLC) procedure

INTERVENTIONS:
Procedure: endoloop mediated cardioplication (ECLC) procedure — The ECLC surgery first incises the mucosa and submucosa on the small curvature side and posterior side (approximately 3/4 of the total circumference) of the diaphragm level cardia until smooth muscle fibers are exposed; Fix the metal clip covered with nylon rope on the exposed smooth muscle layer, and finally tighten the nylon rope to achieve full folding of the cardia. After the surgery, the patient fasted overnight and received intravenous PPI treatment. On the second day after surgery, a fluid diet was restored and discharge was possible. ECLC is simple, easy to operate, relatively inexpensive, and minimally invasive, and is expected to become a new method for treating severe gastroesophageal reflux disease.

SUMMARY:
Endoscopic full-thickness plication (EFTP) of cardia/fundus has been shown effective in treating GERD patients. However, EFTP requires proprietary equipment that are not available in many countries. Here, we designed a metal clip and endoloop mediated cardioplication (ECLC) procedure to achieve EFTP.

DETAILED DESCRIPTION:
Endoscopic full thickness pancreatography (EFTP) is a minimally invasive surgical method that has emerged in recent years for the treatment of severe gastroesophageal reflux disease. This surgery requires the use of disposable patented instruments, which is expensive and has not entered the domestic market. To this end, we have innovatively developed an endoloop mediated cardioplication (ECLC) that only requires metal clips and nylon ropes. The most common and inexpensive endoscopic consumables can achieve the effect of tightening the lower esophageal sphincter, which is expected to be used for the treatment of gastroesophageal reflux disease. The ECLC surgery first incises the mucosa and submucosa on the small curvature side and posterior side (approximately 3/4 of the total circumference) of the diaphragm level cardia until smooth muscle fibers are exposed; Fix the metal clip covered with nylon rope on the exposed smooth muscle layer, and finally tighten the nylon rope to achieve full folding of the cardia. After the surgery, the patient fasted overnight and received intravenous PPI treatment. On the second day after surgery, a fluid diet was restored and discharge was possible. ECLC is simple, easy to operate, relatively inexpensive, and minimally invasive, and is expected to become a new method for treating severe gastroesophageal reflux disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years old
* hiatal hernia ≤ 3cm
* Sliding hernia ≤ 3cm
* Classic reflux symptoms (heartburn, reflux) lasting for more than 6 months
* Daily PPIs ≥ 6 months
* Esophagitis (Los Angeles grade) Grade A, B, and C
* Gastroesophageal valve I-III grade (Hill grade)
* Pathological esophageal acid exposure (percentage of time with 24-hour esophageal PH<4 <4.2%)
* Normal or near normal esophageal movement (through manometry or impedance)
* The lower esophageal sphincter pressure (LESP) is between 5-15mmHg
* DeMeester score ≥ 14.7 or total reflux episodes>73
* Patients who sign an informed consent form and voluntarily accept surgical expenses.

Exclusion Criteria:

* BMI>35kg/m2
* ASA >II
* Barrett's esophagus
* Hill IV level
* Large esophageal hiatal hernia>3cm
* Esophagitis (Los Angeles grade) Grade D
* Peptic ulcer
* Primary esophageal motility disorders such as achalasia
* Previous esophageal or gastric surgery
* Uncontrolled systemic diseases
* Pregnancy or planned pregnancy within 1 year
* Have a history of cervical fusion surgery, esophageal diverticulum, scleroderma or dermatomyositis, eosinophilic esophagitis, liver cirrhosis or coagulation dysfunction, immune system diseases
* Patients deemed unsuitable for inclusion by researchers.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-12-10 (Estimated); Primary Completion 2024-12-10 (Estimated); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
The total score of the GERD-HRQL questionnaire | at 3 month follow- up
  Questionnaire (GERD-HRQL) : Total Score: Calculated by summing the individual scores toquestions 1-15 Greatest possible score ( worst symptoms)= 75 Lowest possible score ( no symptoms)= 0 Heartburn Score: Calculated by summing the individual scores to questions 1-6 . Worst heartburn symptoms = 30 No heartburn symptoms= 0 Scores of ≤ 12 with each individual question not exceeding 2 indicate heartburn elimination. Regurgitation Score: Calculated by summing the individual scores to questions10-15. Worst regurgitation symptoms = 30 No regurgitation symptoms = 0 Scores of ≤ 12 with each individual question not exceeding 2 indicate regurgitation elimination.

SECONDARY OUTCOMES:
PPI usage | at 3, 6 and 12 month follow- up
  Requirement of PPI for control of symptoms at 3, 6 and 12 months Heartburn and Regurgitation questionnaire 0 =No symptom 1 =Symptoms noticeablebut not bothersome 2=S ymptoms noticeableand bothersome but noteve ry day 3 =Symptoms bothersome every day 4 =Symptoms affect daily activity 5 =Symptoms are incapacitating to do daily activities
Total score of GERD GerdQ questionnaire | at 3 month follow- up
  Questionnaire (GERD-GerdQ ) : Recall the frequency of burning sensation (heartburn) after your sternum in the past 7 days;How often do you feel stomach contents (liquid or food) returning to your throat or mouth (reflux) in the past 7 days?How often did you feel pain in the center of your upper abdomen in the past 7 days?How often did you feel nauseous in the past 7 days?How often have you had difficulty getting good night sleep due to heartburn and/or reflux in the past 7 days? Looking back on the past 7 days, in addition to the medication advised by the doctor, did you take additional medication to alleviate the frequency of heartburn and/or reflux? (such as calcium carbonate, aluminum hydroxide, and other antacids).0 days are 0 points, 1 day is 1 point, 2-3 days are 2 points, and 4-7 days are 3 points. Add up the scores for each item to obtain the total score.
Total score of GERD GerdQ and GERD HRQL questionnaires | at 6 and 12 month follow- up
  as mentioned above
Esophageal acid reflux and DeMeester score | at 3, 6, and 12 months follow- up
  There are three monitoring indicators: (1) Total acid exposure time: percentage of total time with pH<4 in 24 hours, standing and lying positions; (2) Acid exposure frequency: number of times with pH<4; (3) Duration of acid exposure: number of times with reflux duration ≥ 5 minutes and maximum reflux duration. The above indicators were calculated using the Demester system of the computer to obtain the total score. Foreign data suggests a normal value of<14.72, while limited domestic data suggests a value of<12.4. The normal 24-hour esophageal pH reference value is: the total time for pH<4 is<4%, the number of reflux times within 5 minutes is ≤ 2, and the longest reflux duration is<16 minutes.
Healing status of reflux esophagitis and damaged mucosa | at 3, 6, and 12 months
  Repair of esophageal mucosa at the surgical site
Safety evaluation indicators | at 0, 3, 6, and 12 months
  The incidence of intraoperative and postoperative bleeding and perforation; Postoperative pain score

IPD SHARING:
Plan to Share IPD: No